CLINICAL TRIAL: NCT02163252
Title: Does Early Intervention Improve Weight Loss Outcomes Among Individuals Enrolled in an Internet-based Weight Loss Program?
Brief Title: Using a State-wide Initiative to Disseminate Effective Behavioral Weight Loss Strategies: Study 5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Jessica Unick, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211699_5
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): A 12-week internet-based weight loss program that involves weekly video lessons, a self-monitoring platform where participants submit their weight, calorie, and activity information, and weekly automated feedback.
  Interventions: Behavioral: Standard
- Early intervention (Experimental): Participants randomized to Early Intervention will receive the same internet-based weight loss program compared to the Standard group. In addition, Early Intervention participants achieving less than optimal weight loss following several weeks of treatment will be given the opportunity to come to the Weight Control and Diabetes Research Center for an individual visit. At this visit, an interventionist will discuss with the participant any barriers that he or she may be experiencing and recommend alternate strategies to assist in their weight loss. One such strategy would be to recommend the use of meal replacement products or portion controlled meals. In addition to this one-time visit, the interventionist will follow up with the participant via phone weekly, for 2 weeks following this in-person visit.
  Interventions: Behavioral: Early Intervention

INTERVENTIONS:
Behavioral: Standard
  Arms: Standard
Behavioral: Early Intervention
  Arms: Early intervention

SUMMARY:
The purpose of this study is to examine whether providing additional intervention support to individuals with lower than expected weight loss within the initial stages of an internet-based behavioral weight loss program improves weight loss outcomes at Week 12, compared to the internet program alone.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* BMI >=25 kg/m2
* No health problems that make weight loss or unsupervised exercise unsafe
* English speaking
* Access to computer/internet

Exclusion Criteria:

* report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire 62 (PAR-Q; items 1-4).
* Individuals endorsing joint problems, prescription medication use or other medical conditions that could limit exercise will be required to obtain written consent to participate from a health care provider
* are currently pregnant or intend to become pregnant in the next 12 months
* are planning to move outside of the state within the next 4 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in weight | 12-week

SECONDARY OUTCOMES:
frequency of self-monitoring | 12 weeks
  A secondary aim is to examine whether the provision of additional intervention support improves the frequency of self-monitoring as measured by the number of days that an individual logged their calorie information on the study website.
exercise minutes | 12 weeks
  A secondary aim is to examine whether the provision of additional intervention support improves the number of exercise minutes reported each week, as logged by the individual on the study website.

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States